CLINICAL TRIAL: NCT04928417
Title: Exacerbations and Their Outcomes International (EXACOS International): Understanding Burden of Severe Exacerbations of COPD and Association Between Frequency of Severe Exacerbations Clinical and Health-care Utilization Outcomes in Less Well-resourced Countries
Brief Title: Exacerbations and Their Outcomes International (EXACOS International)
Acronym: EXACOS-Intl
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00042
Record Dates: First submitted 2021-06-10; First posted 2021-06-16 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, cross-sectional study with retrospective data collection from medical records. During the cross-sectional study visit, data will be captured through the use of electronic Case Report Forms (eCRFs). As there will be only one study visit, no prospective data collection will take place, nor collection of data that are not part of the routine clinic visit.

For understanding the burden of severe exacerbations of COPD and the association between frequency of severe exacerbations and clinical and health-care utilization outcomes in less well-resourced countries

DETAILED DESCRIPTION:
Observational, cross-sectional study with retrospective data collection from medical records. During the cross-sectional study visit, data will be captured through the use of electronic Case Report Forms (eCRFs). As there will be only one study visit, no prospective data collection will take place, nor collection of data that are not part of the routine clinic visit.

For understanding the burden of severe exacerbations of COPD and the association between frequency of severe exacerbations and clinical and health-care utilization outcomes in less well-resourced countries

Patients, treated by pulmonologists, with an investigator-confirmed diagnosis of COPD for at least 5 years from the index date (the date that signed Informed Consent was obtained) and who meet all of the inclusion and none of the exclusion criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they meet the following inclusion criteria:

  1. have an investigator-confirmed diagnosis of COPD of at least 5 years and are over the age of 40 years old;
  2. are smokers or ex-smokers (quit smoking no longer than 15 years before the study visit);
  3. have COPD-related data recorded in (electronic) medical records for at least 5 years, including spirometry and medication data;
  4. have signed a written Informed Consent Form

Exclusion Criteria:

* Patients will be excluded from participation if they meet any of the following exclusion criteria:

  1. have a diagnosis of bronchiectasis, sarcoidosis, Interstitial Lung Diseases, or Idiopathic pulmonary fibrosis. This is because differentiating deteriorations in symptoms/exacerbations in these individuals at attributing them to COPD is impossible

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, treated by pulmonologists, with an investigator-confirmed diagnosis of COPD for at least 5 years from the index date (the date that signed Informed Consent was obtained) and who meet all of the inclusion and none of the exclusion criteria detailed below will be included.
Sampling Method: Probability Sample
Enrollment: 1762 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Estimate the frequency of severe Acute exacerbation of COPD, in a COPD population | 5 YEAR
  Number of severe Acute exacerbation of COPD events and interval between severe AECOPDs over the past 5 years
c) To describe lung function decline over time (FEV1) | 5 YEAR
  At least 2 (Forced expiratory volume in 1 second)FEV1 measurements at least 6 months apart
Health care resource utilization in AECOPD | 5 YEARS
  Number of hospitalizations due to AECOPD in 60 months prior to study visit and time between hospitalizations

SECONDARY OUTCOMES:
Modified Medical Research Council (mMRC) dyspnea scale measured at time of the visit | 1 YEAR
  Modified Medical Research Council (mMRC) dyspnea questionnaire to asses the grade as follow:
  * Grade 0: I only get breathless with strenuous exercise
  * Grade 1: I get short of breath when hurrying on the level or walking up a slight hill
  * Grade 2: I walk slower than people of the same age on the level because of breathlessness, or I have to stop for breath when walking on my own pace on the level
  * Grade 3: I stop for breath after walking about 100 meters or after a few minutes on the level
  * Grade 4: I am too breathless to leave the house or I am breathless when dressing or undressing

CONTACTS AND LOCATIONS:
Locations (18):
- Research Site, Santiago, Chile
- Mexico (2):
  - Research Site, Guadalajara
  - Research Site, Puebla City
- Russia (9):
  - Research Site, Blagoveshchensk, Russia
  - Research Site, Chelyabinsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Voronezh
  - Research Site, Yekaterinburg
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: EXACOS_CSR_Synopsis_Final_03Oct2023.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00042&attachmentIdentifier=f9291549-0d9b-48a2-aa09-f406019af05d&fileName=EXACOS_CSR_Synopsis_Final_03Oct2023.pdf&versionIdentifier=